CLINICAL TRIAL: NCT02711085
Title: The Systematic Merging of Biology, Mental Health and Environment (SYMBIOME) Longitudinal Databanking Project
Brief Title: Modeling Post-traumatic Pain and Recovery: The SYMBIOME Longitudinal Cohort Study
Acronym: SYMBIOME
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Canadian Pain Society (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 106140
Record Dates: First submitted 2015-12-16; First posted 2016-03-17 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2018-12

CONDITIONS: Musculoskeletal Pain; Injuries
MeSH Terms: conditions — Musculoskeletal Pain; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Saliva Blood Hair Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute trauma: Those within the first 3 weeks of a non-catastrophic injury affecting the musculoskeletal system, including but not limited to whiplash or other road-traffic collisions, sports injuries, work-related injuries, sprains, strains, slips and falls and non-displaced fractures that don't require surgical correction.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention - observational study

SUMMARY:
This study will explore the contribution of stress-system activity to pain and functional disability in the acute stage of traumatic musculoskeletal injury, and to the maintenance of symptoms after 3, 6 and 12 months post-injury.

DETAILED DESCRIPTION:
Purpose: The purpose of this protocol is to establish a longitudinal database of data collected from people having experienced an acute traumatic injury to their musculoskeletal system. This includes injuries commonly considered 'non-catastrophic' or 'minor' soft tissue injuries such as whiplash, low back injuries, sports or slip and fall-type injuries that result in sprain/strain of muscle, tendon, ligament or other such soft tissues. Uncomplicated bony fractures (those that are managed through casting only, non-surgical) will also comprise this cohort. The data will include biological specimens, psychological and cognitive profiles, and social/environmental indicators. This protocol represents the start of the SYStematic Merging of Biology, Mental health and Environment (SYMBIOME) project from the emerging Solving Traumatic pain and disability through Advanced Research Translation (START) research group centred at Western. Over time, this database will allow rich exploration of complex interactions between biology, psychology and environment as they relate to the resolution of traumatic pain and disability, or similarly the persistence thereof. Additional research ethics board (REB) applications will be submitted as those projects are ready to be formally conducted.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants:

1. Will be aged 18 years or older
2. Will be able to speak and understand conversational (grade 6) English
3. Will be free of cognitive impairments that would interfere with ability to follow directions (e.g. diagnosed Alzheimer's Dementia, Down's Syndrome)
4. Will be free of neuromuscular disorder that impairs mobility (e.g. stroke, multiple sclerosis, cerebral palsy, ALS)
5. Will be free of active malignancies for the past 5 years
6. Will be free of systemic inflammatory conditions, including rheumatoid or psoriatic arthritis, scleroderma, or systemic lupus erythematosus
7. Will not have been diagnosed with a concussion over the previous 6 months (including the current injury)
8. Will not have been hospitalized overnight over the previous 6 months (including the current injury)
9. Will not have taken steroid-based medications (either prescribed or self-administered) over the previous 6 months
10. Will not have required surgical correction/relocation as a result of the trauma (e.g. open reduction/internal fixation of a fracture). -

Exclusion Criteria:

* Those who are under the influence of drugs or alcohol, or are otherwise not able to provide appropriate informed consent at the time of contact and those with no fixed address will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 or over presenting for issues of pain/limited function arising from acute (<3 weeks) injury affecting the musculoskeletal system that does not require hospital admission or surgery ('minor' injuries).
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Recovery change | 1, 2, 3, 6, and 12 months
  Change in Satisfaction and Recovery Index
Functional Recovery | 1, 2, 3, 6, 12 months
  Brief Pain Inventory - Interference Subscale

SECONDARY OUTCOMES:
Change in Work status | 1, 2, 3, 6, and 12 months
  Work status in relation to pre-injury status
Change in Pain | 1, 2, 3, 6, and 12 months
  Numeric Rating Scale
Change in Post-traumatic Stress | 1, 2, 3, 6, and 12 months
  PTSD Checklist
Change in Depressive Symptoms | 1, 2, 3, 6, and 12 months
  Patient Health Questionnaire - 9

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified database will be made available on a cost-recovery basis as data accrue.

REFERENCES:
- [Derived] Modarresi S, MacDermid JC, Suh N, Elliott JM, Walton DM. How Is the Probability of Reporting Various Levels of Pain 12 Months After Noncatastrophic Injuries Associated with the Level of Peritraumatic Distress? Clin Orthop Relat Res. 2022 Feb 1;480(2):226-234. doi: 10.1097/CORR.0000000000002024. PMID 34705736
- [Derived] Lee JY, Fakhereddin M, MacDermid JC, Elliott JM, Schabrun SM, Walton DM. An Exploration of Blood MarkerxEnvironment Interaction Effects on Pain Severity and Interference Scores in People With Acute Musculoskeletal Trauma. Clin J Pain. 2021 Oct 1;37(10):747-758. doi: 10.1097/AJP.0000000000000961. PMID 34292185
- [Derived] Ghodrati M, Walton DM, MacDermid JC. Exploring the Domains of Gender as Measured by a New Gender, Pain and Expectations Scale. Womens Health Rep (New Rochelle). 2021 Apr 9;2(1):87-96. doi: 10.1089/whr.2020.0109. eCollection 2021. PMID 33937906
- [Derived] Lee JY, Walton DM, Tremblay P, May C, Millard W, Elliott JM, MacDermid JC. Defining pain and interference recovery trajectories after acute non-catastrophic musculoskeletal trauma through growth mixture modeling. BMC Musculoskelet Disord. 2020 Sep 17;21(1):615. doi: 10.1186/s12891-020-03621-7. PMID 32943021